CLINICAL TRIAL: NCT06161220
Title: A Three-Way Crossover Thorough QT/QTc Study to Evaluate the Electrocardiographic Effects of a Supratherapeutic Dose of Carbidopa in Healthy Subjects
Brief Title: A TQT Study to Evaluate the Electrocardiographic Effects of Carbidopa in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Impax Laboratories, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IPX203-102-23
Record Dates: First submitted 2023-11-30; First posted 2023-12-07 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Cardiac Repolarization in Healthy Subjects
MeSH Terms: interventions — Carbidopa

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blinded (for test and negative control) and open label (for active control)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Carbidopa capsule (Experimental): Dose: 4x 100 mg
  Interventions: Drug: Carbidopa capsule; Drug: Moxifloxacin Tablets, USP; Drug: Placebo
- Moxifloxacin Tablets, USP (Active Comparator): Dose: 400 mg
  Interventions: Drug: Carbidopa capsule; Drug: Moxifloxacin Tablets, USP; Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Carbidopa capsule; Drug: Moxifloxacin Tablets, USP; Drug: Placebo

INTERVENTIONS:
Drug: Carbidopa capsule — Dose: 4x 100 mg
Drug: Moxifloxacin Tablets, USP — Dose: 400 mg
Drug: Placebo — Placebo capsules matching the carbidopa capsules

SUMMARY:
The purpose of this trial is to assess the effects of a single supratherapeutic dose of carbidopa on cardiac repolarization relative to placebo in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females aged 18 to 55 years (both inclusive)
* For female subjects of childbearing potential, use of double contraception method
* Body Mass Index (BMI) 18.5 to <30 kg/m² at Screening, with a minimum weight of 55kg
* Subject with no clinically significant abnormal serum biochemistry, hematology and urine examination values at screening
* Subject with negative urine screen for drugs of abuse at screening
* Subject with negative human immunodeficiency virus (HIV), hepatitis B surface antigen (Hep B) and hepatitis C virus antibody (Hep C) results at screening
* Subject must be willing to communicate with the investigator and site staff and comply with all study procedures and requirements
* Subject must be able to provide written, informed consent including compliance with the requirements listed in the consent form
* Subject must be able and willing to swallow whole capsules without breaking, cutting, or chewing

Exclusion Criteria:

* History or presence of systemic diseases at Screening, which as judged by the investigator, may affect the outcome of this study, include, but not limited to significant: cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Female subjects who are pregnant or lactating
* Knowledge of any kind of cardiovascular disorder/condition known to increase the possibility of QT prolongation or history of additional risk factors for Torsade de Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome or Brugada Syndrome) or cardiac conduction disorders
* Resting supine heart rate less than 50 beats per minute or greater than 100 beats per minute
* Resting supine systolic blood pressure less than 90 mmHg or greater than 140 mmHg; resting supine diastolic blood pressure less than 50 mmHg or greater than 90 mmHg.
* Clinically significant (as determined by the Investigator) ECG abnormalities at Screening, including:

  1. QTcF > 450 ms for female and >430 ms for male
  2. QRS > 110 ms
  3. PR > 200 ms
  4. QTcF > 450 ms for female and >430 for male
  5. QRS > 110 ms
  6. PR > 200 ms
  7. Resting supine HR <50 beats per minute (bpm) or >100 bpm (may be repeated once at the discretion of the investigator)
  8. Second or third-degree AV block
  9. Any rhythm other than sinus rhythm, which is interpreted by the Investigator to be clinically significant
  10. Bundle Branch Block
  11. premature atrial and ventricular contractions,
  12. nonspecific T-wave changes
* Positive urine/serum drug screen at Screening or Day -1 for each Period
* History of significant alcohol abuse or drug abuse within one year prior to Screening.
* Use of prescription medication (with the exception of medically approved hormonal contraceptives) including MAO inhibitors in the 30 days prior to admission into Period 1 and over-the-counter medications including vaccines, vitamins, and herbal remedies within 14 days prior to admission of Period 1 till completion of the study (EOS or ET)
* History of unexplained loss of consciousness, unexplained syncope, unexplained irregular heartbeats or palpitations or near drowning with hospital admission
* Subjects who received any investigational drug within the longer of 30 days or 5 half-lives of Day 1 dosing of SM
* Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study
* Use of medications in the 90 days before admission of the study that are known to prolong the QT/QTc interval.
* Family history of QTc prolongation or of unexplainable sudden death at <50 years of age. For this study, family is defined as 1st degree relative (i.e., mother, father, siblings, children) or 2nd degree relative (grandparents, grandchildren, half-siblings, aunt/uncle, niece/nephew).
* Subjects who cannot refrain from using tobacco of any kind within 30 days prior to admission (Day -1) of Period 1 until the last blood sample collection of study
* Subjects who cannot refrain from consumption of alcohol or alcohol containing products or xanthine-containing foods or beverages (like chocolate, tea, coffee or cola drinks) within 48 hours prior to admission (Day -1) of Period 1 till the last blood sample collection of study
* Subjects who participate in other drug research study during the study.
* Subjects who cannot refrain from donating blood or plasma for 30 days and 14 days (respectively) prior to dosing, during the study, and for at least 4 weeks after completing the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2023-12-03 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline QTcF (ΔQTcF) | Predose to 24 hours postdose
  Change-from-baseline QTcF ( QTcF) will allow evaluation of the effects of carbidopa and moxifloxacin on cardiac repolarization based on model derived placebo-corrected ΔQTcF (ΔΔQTcF).

SECONDARY OUTCOMES:
Change from baseline HR, PR, and QRS | Predose to 24 hours postdose
  Change from baseline HR, PR, and QRS (ΔHR, ΔPR, ΔQRS) will also be measured to allow evaluation of the effects of carbidopa and moxifloxacin on other ECG parameters based on model derived placebo-corrected ΔHR, ΔPR, and ΔQRS (ΔΔHR, ΔΔPR, and ΔΔQRS).

CONTACTS AND LOCATIONS:
Locations (1):
- AXIS Clinicals, LLC, Dilworth, Minnesota, United States